CLINICAL TRIAL: NCT05585424
Title: Effectiveness of a Program Based on Observation-action Training (AOT) on Motor, Functional and Cognitive Aspects in Patients With Cognitive Impairment.
Brief Title: Effectiveness of a Program Based on Observation-action Training (AOT) in Patients With Cognitive Impairment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Estrada Barranco, PhD in health sciences, Universidad Europea de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cecilia Estrada Barranco
Record Dates: First submitted 2022-10-11; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Cognitive Impairments
Keywords: Action observation treatment; Cognitive impairment; Mirror neurons; Elderly people
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: nonranzomized controlled trial study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients in the experimental group were paired so that each patient with MCI faced a patient with ModCI. During the sessions, two therapists performed the upper limb activities that only the MCI patients could see and they performed them by imitation
  Interventions: Other: AOT intervention
- Control group (No Intervention): The CG was assessed at baseline and after one month and continued with their usual activities in the nursing home.

INTERVENTIONS:
Other: AOT intervention — The treatment will last 4 weeks, with an intensity of 3 sessions per week. During the sessions the MCI patient will observe his MCI partner and perform a programme of upper limb motor activities. At the same time the mild patient imitates the movement performed by the physiotherapist, all based on the AOT.
  The activities will be based on items of the FUGL-MEYER scale. The sessions will last between 15 and 20 minutes and will be held three days a week. The intervention will last 5 weeks, with an initial assessment, 11 intervention sessions and a final assessment.
  Arms: Experimental Group

SUMMARY:
The objective of this study is to assess motor and social interaction changes after AOT intervention in patients with mild cognitive impairment and Moderate cognitive impairment.

The planned sample size is 11 pairs in the experimental group and 11 pairs in the control group. Each group will be composed of eleven subjects with moderate cognitive impairment (MCI) and eleven with mild cognitive impairment (MCI), assessed by the minimental test. During the sessions, the MCI patient will observe his MCI partner and perform a programme of motor activities for the upper limb. At the same time the mild patient imitates the movement performed by the physiotherapist, all based on the AOT.

The activities will be based on items of the FUGL-MEYER scale. Data will be collected at the functional level, with respect to motor changes and also social modifications that have been perceived by the participants, carers and therapists.

The variables considered in this study are, as primary variables, motor changes, using the Fugl-Meyer scale, and perception with respect to social interaction; as well as mood. The latter two will be collected through interviews with patients, caregivers and therapists.

The impact on patient independence (Barthel index score) will also be considered. Finally, data will be analysed using SPSS statistical software. Non-parametric tests for related samples will be used in order to study changes in the variables collected before and after the intervention. The sample will be recruited from the old people's home "Nuestra Señora de la Soledad" in Parla, Madrid (collaboration agreement attached) depending on whether or not they meet the inclusion criteria.

DETAILED DESCRIPTION:
Previous work has demonstrated the effectiveness of observational learning. A previous study on children with cerebral palsy "Efficacy of a home-based platform for child-to-child interaction on hand motor function in unilateral cerebral palsy" presented by Naura, Avanzini, Rizzolatti and Fabbri-Destro, showed that motor learning by observation is greater and presents more evident benefits when subjects learn from other patients with the same condition and less severity than when they learn by observing the therapist or another person without motor impairment. This work seeks to measure the improvements, both motor, functional and social, that patients with cognitive impairment can achieve with such an intervention.

This work is an experimental study based on the stimulation of mirror neurons. The planned sample size is 11 pairs in the experimental group and 11 pairs in the control group. Each group will be composed of eleven subjects with moderate cognitive impairment (MCI) and eleven with mild cognitive impairment (MCI), assessed by the minimental test. During the sessions, the MCI patient will observe his MCI partner and perform a programme of motor activities for the upper limb. At the same time the mild patient imitates the movement performed by the physiotherapist, all based on the AOT.

The activities will be based on items of the FUGL-MEYER scale. The sessions will last between 15 and 20 minutes and will be held three days a week. The intervention will last 5 weeks, with an initial assessment, 11 intervention sessions and a final assessment.

Inclusion criteria are: institutionalised patients over 65 years of age with mild cognitive impairment (minimental test between 19 and 23) or moderate cognitive impairment (minimental test 14-18); patients who perform physiotherapy exercises twice a week or attend occupational therapy twice a week; patients supervised by geriatric assistants or nurses during basic activities of daily living.

Exclusion criteria are considered to be: patients with musculoskeletal and neuro-musculoskeletal pathology of the dominant upper limb (outside MCI and MCI); presentation of visual deficit not correctable with glasses; patients with aggressive behavioural alterations or emotional lability; presentation of severe hypoacusis not correctable with hearing aids.

Data will be collected at the functional level, with respect to motor changes and also social modifications that have been perceived by the participants, carers and therapists.

The variables considered in this study are, as primary variables, motor changes, using the Fugl-Meyer scale, and perception with respect to social interaction; as well as mood. The latter two will be collected through interviews with patients, caregivers and therapists.

As secondary variables, functional changes in feeding (feeding time, errors in food intake, accuracy in bringing food to the mouth) will be considered. The impact on patient independence (Barthel index score) will also be considered. Finally, data will be analysed using SPSS statistical software. Non-parametric tests for related samples will be used in order to study changes in the variables collected before and after the intervention. The sample will be recruited from the old people's home "Nuestra Señora de la Soledad" in Parla, Madrid (collaboration agreement attached) depending on whether or not they meet the inclusion criteria.

Participants and/or legal representatives will sign an informed consent form once they have decided to participate after having received an information sheet with a detailed description of the study procedure and clarification of any doubts they may have (attached below). A consent form for the recording of patients during the assessments is also attached. The patient's personal data are coded in order to maintain their anonymity.

The handling and confidentiality of the data will be carried out in accordance with the regulations in force and following the Organic Law 3/2018, on the Protection of Personal Data and guarantee of digital rights.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalised patients over 65 years of age.
* Mild cognitive impairment (minimental test between 19 and 23) or moderate cognitive impairment (minimental test 14-18);
* Patients supervised by geriatric or nursing assistants during basic activities of daily living

Exclusion Criteria:

* Patients with musculoskeletal and neuro-musculoskeletal pathology of the dominant upper limb (outside MCI and MCI);
* Presentation of visual deficit not correctable with glasses;
* Patient with aggressive behavioural disturbance or emotional lability;
* Patient with severe hypoacusis not correctable with hearing aids.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Upper limb functionality measured with upper limb subsection of the Fugl Meyer scale | one month
  The upper limb subsection has 33 items, with the maximum score of 66 being associated with the best upper limb motor function and 0 being the minimum score
Independence in activities of daily living measured with Barthel Índex | one month
  here are 10 items that add up to 5 or 10 points and total up to a maximum of 100 when the person is independent in BADLs
Cognitive impairment measured with Mini-Mental State Examination (MMSE) | one month
  The MMSE assesses different cognitive functions (orientation, memory, attention and calculation, language, construction, praxis and reasoning). The maximum score is 30. A score of 23 or lower is associated with cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Estrada Barranco, Dra, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Cecilia Estrada Barranco, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No